CLINICAL TRIAL: NCT05003596
Title: Efficacy of Steroids on Functional Outcomes After Musculoskeletal Injuries of the Hand
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Robert Wood Johnson Barnabas Health (Other)
Collaborators: Brielle Orthopedics (Unknown); University Orthopedics Associates (Unknown)
Responsible Party: Principal Investigator, Bobby Varghese, Co-Investigator, Robert Wood Johnson Barnabas Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2021000732
Record Dates: First submitted 2021-07-28; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Hand Injuries; Finger Injuries
MeSH Terms: conditions — Hand Injuries; Finger Injuries | interventions — Methylprednisolone; Acetaminophen; Narcotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: data without intervention identification will be analyzed by outcome assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Steroid Group (Experimental): Patients receive 21 tablets of 4 mg methylprednisolone to be taken by mouth over a 6 week taper. Patients will be advised to not take other anti-inflammatory medications like NSAIDs.
  Interventions: Drug: Methylprednisolone Tablet
- Control Group (Active Comparator): Patients will recieve standard treatment that focuses on mobilization and stabilization using common techniques like buddy taping and splinting. Pain control will be managed using non-NSAID medications like Tylenol or opioid narcotics when deemed medically necessary.
  Interventions: Other: Standard Mobilization Treatment

INTERVENTIONS:
Drug: Methylprednisolone Tablet — Subjects will take a quantity 21 4mg tablets over a 6 week taper.
  Other Names: Solu-Medrol Dosepak
  Arms: Steroid Group
Other: Standard Mobilization Treatment — standard treatment of hand injuries with focus on mobilization. No anti-inflammatory medications. Pain management via Tylenol or narcotics if deemed necessary.
  Other Names: buddy taping; finger splint; tylenol; narcotics
  Arms: Control Group

SUMMARY:
Steroids are often prescribed for their anti-inflammatory effects in patients with musculoskeletal injuries. Studies have shown that steroids may reduce pain and swelling, but their effects on range of motion and functional outcomes have not been illustrated. With this study, we aim to evaluate the effect of steroids on range of motion and functional outcomes in non-operatively managed musculoskeletal injuries of the hand.

DETAILED DESCRIPTION:
Previous studies have investigated the effect of steroids on bone healing, edema reduction and postoperative pain. However, there seems to be a lack of literature on whether the use of steroids for their anti-inflammatory effects actually lead to improved range of motion and functional capacity. If the data shows that steroids do indeed help patients achieve increased functional outcomes, they may be used with higher confidence in their beneficial contribution to patient treatment and quality of life. If, however, the data show that steroids do not confer a significant benefit, they can be disregarded as they will avoid the risks associated with steroid use. We aim to investigate if the use of methylprednisolone will result in significantly improved ranges of motion and self-reported function compared to a control group at each measurement time point.

ELIGIBILITY:
Inclusion Criteria:

* Patients with soft tissue injuries and stable fractures from the metacarpophalangeal joint to the distal phalanx

Exclusion Criteria:

* Patients at increased risk of serious side effects of steroid administration.
* Patients unable to provide consent
* Unable to swallow oral medications
* Pregnant women
* ages less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
wrist flexion | initial
  degrees of wrist flexion
wrist flexion | 3 weeks
  degrees of wrist flexion
wrist flexion | 6 weeks
  degrees of wrist flexion
wrist flexion | 12 weeks
  degrees of wrist flexion
wrist extension | 12 weeks
  degrees of wrist extension
wrist extension | 6 weeks
  degrees of wrist extension
wrist extension | 3 weeks
  degrees of wrist extension
wrist extension | initial
  degrees of wrist extension
hand supination | initial
  degrees of hand supination
hand supination | 3 weeks
  degrees of hand supination
hand supination | 6 weeks
  degrees of hand supination
hand supination | 12 weeks
  degrees of hand supination
hand pronation | initial
  degrees of hand pronation
hand pronation | 3 weeks
  degrees of hand pronation
hand pronation | 6 weeks
  degrees of hand pronation
hand pronation | 12 weeks
  degrees of hand pronation
wrist ulnar deviation | initial
  degrees of wrist ulnar deviance
wrist ulnar deviation | 3 weeks
  degrees of wrist ulnar deviance
wrist ulnar deviation | 6 weeks
  degrees of wrist ulnar deviance
wrist ulnar deviation | 12 weeks
  degrees of wrist ulnar deviance
wrist radial deviation | initial
  degrees of radial deviance of the wrist
wrist radial deviation | 3 weeks
  degrees of radial deviance of the wrist
wrist radial deviation | 6 weeks
  degrees of radial deviance of the wrist
wrist radial deviation | 12 weeks
  degrees of radial deviance of the wrist
MCP, DIP, PIP of digits 2-5: Flexion | initial
  degrees of flexion for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: Flexion | 3 weeks
  degrees of flexion for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: Flexion | 6 weeks
  degrees of flexion for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: Flexion | 12 weeks
  degrees of flexion for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: Extension | initial
  degrees of extension for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: Extension | 3 weeks
  degrees of extension for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: Extension | 6 weeks
  degrees of extension for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: Extension | 12 weeks
  degrees of extension for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: abduction | initial
  degrees of abduction for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: abduction | 3 weeks
  degrees of abduction for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: abduction | 6 weeks
  degrees of abduction for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: abduction | 12 weeks
  degrees of abduction for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: adduction | initial
  degrees of adduction for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: adduction | 3 weeks
  degrees of adduction for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: adduction | 6 weeks
  degrees of adduction for MCP, DIP, and PIP of digits 2-5
MCP, DIP, PIP of digits 2-5: adduction | 12 weeks
  degrees of adduction for MCP, DIP, and PIP of digits 2-5
Thumb Opposition at MCP | initial
  degrees of thumb opposition
Thumb Opposition at MCP | 3 weeks
  degrees of thumb opposition
Thumb Opposition at MCP | 6 weeks
  degrees of thumb opposition
Thumb Opposition at MCP | 12 weeks
  degrees of thumb opposition
Thumb extension at IP | initial
  degrees of thumb IP extension
Thumb extension at IP | 3 weeks
  degrees of thumb IP extension
Thumb extension at IP | 6 weeks
  degrees of thumb IP extension
Thumb extension at IP | 12 weeks
  degrees of thumb IP extension
Thumb flexion at IP | initial
  degrees of thumb IP flexion
Thumb flexion at IP | 3 weeks
  degrees of thumb IP flexion
Thumb flexion at IP | 6 weeks
  degrees of thumb IP flexion
Thumb flexion at IP | 12 weeks
  degrees of thumb IP flexion
Quick DASH Questionnaire | 6 weeks
  patient-reported outcome survey that evaluates functionality and patient-perceived disability
Quick DASH Questionnaire | 12 weeks
  patient-reported outcome survey that evaluates functionality and patient-perceived disability

SECONDARY OUTCOMES:
VAS Pain Scale | 3 weeks
  visual analog pain scale
VAS Pain Scale | 6 weeks
  visual analog pain scale
VAS Pain Scale | 12 weeks
  visual analog pain scale
Complications | 3 weeks
  list of adverse events
Complications | 6 weeks
  list of adverse events
Complications | 12 weeks
  list of adverse events
Edema Measurements | 3 weeks
  measurements of noted edema to the study area
Edema Measurements | 6 weeks
  measurements of noted edema to the study area
Edema Measurements | 12 weeks
  measurements of noted edema to the study area

CONTACTS AND LOCATIONS:
Overall Officials: Brian Katt, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - Brielle Orthopedics, Brick, New Jersey
  - University Orthopedics Associates, Somerset, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rytter S, Stilling M, Munk S, Hansen TB. Methylprednisolone reduces pain and decreases knee swelling in the first 24 h after fast-track unicompartmental knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Jan;25(1):284-290. doi: 10.1007/s00167-014-3501-8. Epub 2015 Jan 7. PMID 25564196
- [Background] Yang Z, Lim PPH, Teo SH, Chen H, Qiu H, Pua YH. Association of wrist and forearm range of motion measures with self-reported functional scores amongst patients with distal radius fractures: a longitudinal study. BMC Musculoskelet Disord. 2018 May 11;19(1):142. doi: 10.1186/s12891-018-2065-z. PMID 29747624
- [Background] Troullos ES, Hargreaves KM, Butler DP, Dionne RA. Comparison of nonsteroidal anti-inflammatory drugs, ibuprofen and flurbiprofen, with methylprednisolone and placebo for acute pain, swelling, and trismus. J Oral Maxillofac Surg. 1990 Sep;48(9):945-52. doi: 10.1016/0278-2391(90)90007-o. PMID 2395047
- [Background] Boursinos LA, Karachalios T, Poultsides L, Malizos KN. Do steroids, conventional non-steroidal anti-inflammatory drugs and selective Cox-2 inhibitors adversely affect fracture healing? J Musculoskelet Neuronal Interact. 2009 Jan-Mar;9(1):44-52. PMID 19240368
- See also: Rutgers REDCap server that stores study data — http://redcap.rwjms.rutgers.edu